CLINICAL TRIAL: NCT05251766
Title: Nab-paclitaxel Compared With Docetaxel Combined With Epirubicin and Cyclophosphamide in the Neoadjuvant Chemotherapy Breast Cancer
Brief Title: Nab-paclitaxel Compared With Docetaxel in the Neoadjuvant Chemotherapy Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuli Meng (Other)
Responsible Party: Sponsor-Investigator, Xuli Meng, chief physician, Zhejiang Provincial People's Hospital
Organization: Zhejiang Provincial People's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SRMBCNabP2022
Record Dates: First submitted 2022-01-18; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer; Chemotherapy Effect
MeSH Terms: conditions — Breast Neoplasms | interventions — Taxes; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm1: epirubicin + cyclophosphamide followed by docetaxel (Active Comparator): Epirubicin :90 mg/m2, D1, q3W; Cyclophosphamide :600 mg/m2, D1, q3W; 4 cycles, Follow Docetaxel :75 mg/m2, D1, q3W, 4 cycles
  Interventions: Drug: Docetaxel
- Arm2: epirubicin + cyclophosphamide followed by nab-paclitaxel (Experimental): Epirubicin :90 mg/m2, D1, q3W; Cyclophosphamide :600 mg/m2, D1, q3W; 4 cycles, Follow Nab-paclitaxel :260 mg/m2, d1, q3W; 4 cycles
  Interventions: Drug: Nab paclitaxel
- Arm3: nab-paclitaxel combined with epirubicin + cyclophosphamide (Experimental): Nab-paclitaxel :260 mg/m2, D1, q3W; Epirubicin :90 mg/m2, D1, q3W; Cyclophosphamide :600 mg/m2, D1, q3W; 6 cycles
  Interventions: Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Nab paclitaxel — To analyze and compare the efficacy and safety of epirubicin + cyclophosphamide (EC) followed by docetaxel and EC followed by nab-paclitaxel in neoadjuvant chemotherapy of breast cancer; To analyze and compare the efficacy and safety of nab-paclitaxel combined with epirubicin + cyclophosphamide (EC) chemotherapy regimen in neoadjuvant therapy of breast cancer, so as to provide a new treatment option for patients with HER2-negative breast cancer.
  Other Names: Aiyue(Jiangsu Hengrui Pharmaceuticals Co.)
  Arms: Arm2: epirubicin + cyclophosphamide followed by nab-paclitaxel; Arm3: nab-paclitaxel combined with epirubicin + cyclophosphamide
Drug: Docetaxel — To analyze and compare the efficacy and safety of epirubicin + cyclophosphamide (EC) followed by docetaxel and EC followed by nab-paclitaxel in neoadjuvant chemotherapy of breast cancer; To analyze and compare the efficacy and safety of nab-paclitaxel combined with epirubicin + cyclophosphamide (EC) chemotherapy regimen in neoadjuvant therapy of breast cancer, so as to provide a new treatment option for patients with HER2-negative breast cancer.
  Other Names: Tianlun(Yangzijiang Pharmaceuticals Co.)
  Arms: Arm1: epirubicin + cyclophosphamide followed by docetaxel

SUMMARY:
Comparison of docetaxel and Nab-paclitaxel in neoadjuvant chemotherapy for breast cancer

DETAILED DESCRIPTION:
1. To analyze and compare the efficacy and safety of epirubicin + cyclophosphamide (EC) followed by docetaxel and EC followed by nab-paclitaxel in neoadjuvant chemotherapy of breast cancer; 2. To analyze and compare the efficacy and safety of nab-paclitaxel combined with epirubicin + cyclophosphamide (EC) chemotherapy regimen in neoadjuvant therapy of breast cancer, so as to provide a new treatment option for patients with human epidermal growth factor receptor 2(HER2)-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with age range ≥ 18 years;
2. a single invasive breast cancer conforming to the clinical diagnostic criteria and histologically confirmed.
3. HER2 negative breast cancer, tumor >2 cm, clinical staging conforms to T2-4 phase (defined by immunohistochemistry as 0-1+ or by immunohistochemistry as 2+, without HER2 amplification by Fluorescence in situ hybridization(FISH), chemiluminescent in situ hybridization(CISH) or other amplification tests).
4. Known hormone receptor status (estrogen receptor [ER], progesterone receptor [PR]), known Ki67 value;
5. Eastern Cooperative Oncology Group(ECOG) performance status is 0 or 1;
6. patients have not previously had breast cancer treatment.
7. During the study, be able to comply with outpatient treatment, laboratory monitoring and necessary clinical visits;
8. Subjects have the ability to understand, agree and sign the study informed consent form (ICF) before initiating any protocol related procedures; The subject has the ability to express consent (when applicable);
9. Normal blood, kidney and liver functions (ANC ≥ 1500 / mm3, platelet（PLT）≥ 100000 / mm3, serum creatinine and total bilirubin ≤ 1.5 times of the upper limit of normal, glutamic oxalacetic transaminase(AST) and glutamic-pyruvic transaminase（ALT） ≤ 3 times of the upper limit of normal).

Exclusion Criteria:

1. bilateral invasive breast cancer, metastatic disease or other malignant tumors.
2. Surgical axillary staging surgery was performed within 6 months before entering the study;
3. Pregnant or lactating women; Patients with fertility are unwilling or unable to take effective contraceptive measures;
4. before the start of the study, radiotherapy, chemotherapy, biological therapy and / or hormone therapy for the current diagnosis of breast cancer were carried out.
5. Patients with central nervous system metastasis or > grade 1 peripheral neuropathy;
6. Patients with severe myelosuppression at the time of screening;
7. Patients with severe liver dysfunction (child's class III) or renal dysfunction at the time of screening;
8. Other concomitant diseases that the researchers believe are seriously harmful to the safety of patients or will hinder the implementation or completion of treatment plan (such as untreated congenital heart disease, glomerulonephritis, etc.);
9. Allergic to albumin for injection, paclitaxel, epirubicin, cyclophosphamide and docetaxel;
10. Patients with mental disorders;
11. Subjects who are participating in other clinical studies or whose first medication time is less than 4 weeks (or 5 half lives of the study drug) from the end of the previous clinical study (last administration);
12. Other situations that may affect the progress of clinical research and the judgment of research results and are not suitable for inclusion in the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-20 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response (pCR) rate | 21 weeks
  Proportion of PCR patients in enrolled breast cancer patients

SECONDARY OUTCOMES:
Total clinical response rate | 21 weeks
  The clinical response rate was assessed by ultrasound measurement of tumor size